CLINICAL TRIAL: NCT05997342
Title: A Phase I Clinical Trial to Evaluate the Safety and Tolerability of TQB3912 Tablets in Subjects With Advanced Malignancies
Brief Title: A Clinical Study of TQB3912 Tablets in Patients With Advanced Malignant Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3912-I-01
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignant Neoplasm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3912 tablets (Experimental): TQB3912 tablets, 28 days as a treatment cycle.
  Interventions: Drug: TQB3912 tablets

INTERVENTIONS:
Drug: TQB3912 tablets — TQB3912 is a small molecule Phosphorylated protein kinase inhibitor. Activation of the pathway plays an important role in cell survival, proliferation, migration, and differentiation.

SUMMARY:
This is a study to evaluate the maximum tolerated dose (MTD), occurrence of all adverse events (AEs) and serious adverse events (SAEs), pharmacokinetic parameters and antitumor effect of TQB3912 tablets in Chinese adult patients with advanced malignant neoplasm. The study was divided into phase Ia and phase Ib, Phase Ia: Dose escalation period, to evaluate the safety and tolerability of TQB3912 tablets, determine MTD; Phase Ib: Effectiveness exploration period, to expand the safe and effective dose group, and to recommend appropriate dosage and method for subsequent clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntarily join the study, sign the informed consent form, and have good compliance.
* Aged from 18 to 75 years; Eastern Cooperative Oncology Group performance status score: 0-2; at least 3 months of expected survival period.
* Subjects with relapse advanced malignant solid tumors clearly diagnosed by pathology and/or cytology.
* The function of main organs is normal.
* Subjects need to adopt effective methods of contraception.

Exclusion Criteria:

* Subjects with other malignancies currently or suffered within 3 years.
* Subjects with Grade 1 or above unhealed toxicity reaction of Common Terminology Criteria for Adverse Events Version 5.0 due to previous antitumor treatment.
* Subjects who have received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before first administration.
* Subjects with long lasting wounds or fractures.
* Subjects with a history of psychotropic drug abuse unable to quit or with mental disorders.
* Subjects with any severe and/or uncontrolled disease.
* Subjects who have received surgery, chemotherapy, radiotherapy or other anticancer therapies 4 weeks before the first administration.
* Subjects who have taken Chinese patent medicines with anti-tumor indications in the drug instructions that National Medical Products Administration approved within 2 weeks before the first administration.
* Subjects with pleural effusion, pericardial effusion or ascites that cannot be controlled and need repeated drainage.
* Subjects who have participated in other clinical studies within 4 weeks before the first administration.
* According to the judgment of the investigators, there are accompanying diseases that seriously endanger the safety of patients or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | During the first 28 days.
  Subjects within 28 days after treatment appear the following toxicity reaction relate to the drug: grade III or above of non-hematological toxicity, grade III hematological toxicity, Neutropenia associated with fever.
Maximum tolerated dose (MTD) | During the first 29 days.
  MTD is defined as the highest dosing schedule cohort level at which no more than 1 of 6 patients experience a Dose Limiting Toxicity (DLT).
Overall response rate (ORR) | Up to 2 years
  From the first drug treatment to the last drug treatment.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From the time of informed consent signed to 90 days after the last dose
  Number of patients with adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Incidence of serious adverse events (SAEs) | From the time of informed consent signed to 90 days after the last dose
  Number of patients with serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Disease control rate (DCR) | Up to 2 years
  The proportion of subjects with Complete response (CR), Partial response (PR), or Stable Disease (SD).
Progression-free survival (PFS) | Up to 2 years
  The time from the first dose of TQB3912 to the first occurrence of disease progression or death from any cause.
Duration of Response (DOR) | Up to 2 years
  The time from first documented response to documented disease progression.
Overall survival (OS) | Up to 5 years
  The time between the date of first administration and the date of death due to any cause.
Time to reach maximum (peak) plasma concentration (Tmax) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on single dose; pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQB3912 by assessment of time to reach maximum plasma concentration after single and multiple dosing.
Maximum (peak) plasma drug concentration (Cmax) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on single dose; pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on multiple dose of day 28.
  Cmax is the maximum plasma concentration of TQB3912 or metabolite(s).
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on single dose; pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on multiple dose of day 28.
  Cmax,ss is the maximum steady-state plasma concentration of TQB3912 or metabolite(s).
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on single dose; pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQB3912 by assessment of area under the plasma concentration time curve from the first dose to time t.
Elimination half-life (t1/2) (to be used in one-or non- compartmental model) | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on single dose; pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours after-dose on multiple dose of day 28.
  t1/2 is time it takes for the blood concentration of TQB3912 or metabolite(s) to drop by half.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha, Hunan
  - West China hospital, Sichuan university, Chengdu, Sichuan